CLINICAL TRIAL: NCT00227188
Title: Effectiveness of Prevnar in the Prevention on IPD in the Paediatric Population in Spain
Brief Title: Study Evaluating Prevenar in the Prevention of Invasive Pneumococcal Disease (IPD) in the Paediatric Population in Spain.
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0887-101317
Record Dates: First submitted 2005-09-13; First posted 2005-09-27 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Invasive Pneumococcal Disease
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples without DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Children from 0-5 years of age evaluated for IPD
  Interventions: Drug: Pneumococcal 7-valent conjugate vaccine Prevnar

INTERVENTIONS:
Drug: Pneumococcal 7-valent conjugate vaccine Prevnar
  Other Names: PREVNAR

SUMMARY:
The aim of this study is to evaluate the postlicensure effectiveness of Prevnar in the prevention of IPD in the Spanish paediatric population (children younger than 5 years)

ELIGIBILITY:
Inclusion Criteria:

* All children from 0 up to 5 years attending to the hospital's emergency department will be evaluated for IPD.
* Diagnosis of IPD will be based on positive pneumococcal isolation in any sterile location, such us blood or spinal fluid.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All public and private hospitals with a pediatric department belonging to one of the two autonomous communities.
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2003-05; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Bilbao, Spain

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0887-101317&StudyName=Study%20Evaluating%20Prevenar%20in%20the%20prevention%20of%20invasive%20pneumococcal%20disease%20%20%20%20%28IPD%29%20in%20the%20paediatric%20population%20in%20Spain.